CLINICAL TRIAL: NCT02887079
Title: Research Interest Antiphospholipid in Predicting Embolic Risk During Infective Endocarditis
Acronym: EMBOL-EI
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Christine Selton-Suty, Dr, Central Hospital, Nancy, France
Other Study IDs: PHRCI 2013-13087
Record Dates: First submitted 2016-07-26; First posted 2016-09-01 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Infective Endocarditis
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
EMBOL-EI (Research Interest antiphospholipid antibody for embolic risk prediction in infective endocarditis) is a prospective cohort study with a biological collection.

The main objective is: to re-evaluate the potential value of antiphospholipid (aPL) antibodies as predictors of embolic events in infective endocarditis (IE) in the light of the improved current knowledge on these aPL.

The seconds objectives are: Other plasma biomarkers of hemostasis (coagulation activation markers: D-dimer fragment 1 + 2 of prothrombin; endothelial biomarkers: plasma levels of von Willebrand factor) will be taken into account in the analysis, and interest in predicting embolic risk, alone or in combination with aPL will be investigated.

DETAILED DESCRIPTION:
Criteria of inclusion

* Patient hospitalized in the University Hospital of Nancy with an Endocarditis some as modified Duke criteria by Li.

The patient is eligible if it is considered and treated as a case of infective endocarditis by physicians ensuring its management. The application of the diagnostic classification Duke criteria modified by Li is made after the collection of all the data at the output of the patient. Will be retained for the analysis of patients meeting certain infective endocarditis.

Clinical, microbiological data, derived from complementary therapies and scalable examinations (including the endpoint) were collected during the hospital stay by doctors that support helped a patient technician clinical studies. Each application is reviewed by a multidisciplinary panel of two experts for validation.

Once validated record, the data collection schedule is sent to the Centre d'Investigation Clinique 1433 Epidémiologie Clinique (CIC-EC) to be entered on a database.

A blood sample is taken from each patient at admission. These samples are packaged and stored in a collection. The serum used in search - called anticardiolipin (AC) Immunoglobulin G (IgG) and Immunoglobulin M (IgM) isotype by ELISA.

ELIGIBILITY:
Inclusion Criteria:

* All the patients admitted either in the Infectious Department, in the Cardiology Department or in the Intensive Care Unit of the University Hospital of Nancy and treated for IE.

Exclusion Criteria:

* Patients with a previously known aPL syndrome or illness frequently associated with aPL syndrome (such as lupus)
* Patients with a delay between blood sample and diagnosis of IE longer than 21days
* Patients who had no symptomatic embolic events and no imaging procedure to detect an asymptomatic embolic event

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients admitted either in the Infectious Department, in the Cardiology Department or in the Intensive Care Unit of the University Hospital of Nancy and treated for IE.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Symptomatic or asymptomatic events occurring before and after IE diagnosis | at discharge, an average of 8 weeks after inclusion
  By patients have systematic extra-cardiac imaging

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Besancon, Besançon
  - CHU de Nancy, Nancy

REFERENCES:
- [Result] Selton-Suty C, Maigrat CH, Devignes J, Goehringer F, Erpelding ML, Alla F, Thivilier C, Huttin O, Venner C, Juilliere Y, Doco-Lecompte T, Lecompte T; Endocarditis Team of the University Hospital of Nancy, France. Possible relationship between antiphospholipid antibodies and embolic events in infective endocarditis. Heart. 2018 Mar;104(6):509-516. doi: 10.1136/heartjnl-2017-312359. Epub 2018 Jan 5. PMID 29305562